CLINICAL TRIAL: NCT06044103
Title: Does Adding Patient-controlled Sedation With Propofol During Repair of Obstetric Perineal Lacerations Grade I and II Improve Patient Experiences - a Randomized Control Trial
Brief Title: Patient-controlled Sedation During Repair of Obstetric Perineal Lacerations
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marie Blomberg (Other Government)
Responsible Party: Sponsor-Investigator, Marie Blomberg, Professor in Obstetrics and Gyneacology, Linkoeping University
Organization: Linkoeping University (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PROP(ofol); 2022-502292-39 (EudraCT Number)
Record Dates: First submitted 2023-08-23; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Pain; Patient Satisfaction
Keywords: obstetric perineal lacerations; patient-controlled sedation; propofol
MeSH Terms: conditions — Pain; Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Clinical routine
- Patient-controlled sedation with propofol (Experimental): PCS group
  Interventions: Drug: PDB + PCS

INTERVENTIONS:
Drug: PDB + PCS — Pudendal nerve block (PNB) with ropivacaine AND Patient-controlled sedation with propofol by the participant
  Arms: Patient-controlled sedation with propofol

SUMMARY:
The PROP(ofol)-study (EU CT number: 2022-502292-39-00, protocol number: ) is a clinical trial phase IV single centre prospective randomized controlled trial with parallel groups. A total of 80 women who undergoes examination and repair of obstetric perineal lacerations (grade I and II) are randomized into two arms (1:1); analgesia with pudendal nerve block (PNB) with ropivacaine (clinical routine, control group), or analgesia with PNB in combination with patient-controlled sedation with propofol (PCS, PCS group). The hypothesis is that PNB in combination with PCS improves patient experienced pain/discomfort during the examination and repair of the perineal laceration. The primary endpoint is patient experienced pain/discomfort. Secondary endpoints are time of repairing the perineal laceration, ability to have skin-to-skin contact with the baby during perineal repair, time until micturition after the perineal repair, procedure feasibility, amount of drugs used during perineal repair, and use of pain relief 24h postpartum. The study is planned to start during the second half of 2023 and end during the first half of 2024.

DETAILED DESCRIPTION:
Study design and procedure

1. Study design Clinical trial, Phase IV; therapeutic use. The study is an open prospective randomized controlled low-intervention trial with parallel groups conducted in a clinical unit (single centre). The study will be conducted at the maternity ward, Vrinnevihospital (Norrköping, Sweden), according to the Helsinki Declaration principles.
2. Pre-study visit All patients are informed by about the ongoing study during their last routine visit in full term pregnancy at the out-patientclinic. No informed consent is given at this point.
3. Procedure Standard care are that women with a vaginal delivery undergoes examination, and further repair of perineal laceration after giving birth. Nulliparous women who have given vaginal birth and fulfil the inclusion criteria's will be given verbal and written information about the study. The physician obtains a written informed consent from the participants. Women who fulfil the criteria's and undergoes examination and repair of grades I or II will be included in the study. It shall be noted that no study-related procedures will be done prior signed consent.

   Patients not fulfilling criterions for participation are given standard of care with PNB only.

   Each patient who fulfils participation in the study is allocated consecutively a sealed opaque randomization envelope containing instructions if PNB should be combined with PCS during the procedure or not. There will be two study-arms: pudendal nerve block (group PNB) (todays standard of care) and pudendal nerve block with sedation using PCS with propofol (group PCS). The research subject will be randomized 1:1 to one of the two arms.

   If the research person is randomized to sedation with PCS (group PCS) the midwife or obstetrician, will give additional thorough information and instructions how to operate the PCS device before initiation of the procedure.

   Before PNB is applied, research persons in group PCS is encouraged to start requesting bolus doses from the device until the research person feel comfortable (OAA/S 4/3). During the procedure the midwife may administrate additional local anaesthetics to improve or extend the pain relief as in today's standard care. The procedure takes approximately 30 minutes.

   If the perineal laceration turns out to be of a greater extent, such as perineal laceration grade III-IV during the examination and repairing procedure, the research persons exclude from the study. It is not possible to know if the degree of the perineal laceration is of a larger extent than degree I or II before examination. This is also the routine of today's standard care. The patient will then get today´s standard care with repair of the greater perineal laceration at the operation theatre.

   During and after the procedure the research person is continuously monitored regarding vital signs. Monitoring of vital signs ends when OAA/S 5 is reached after completion of the procedure.

   During and after the procedure the anaesthesiologist is available within minutes if call is made to anaesthesiologist pager.

   Questionnaire regarding patient experiences will be handed out to the research person after the procedure are completed.

   Procedure feasibility is assessed by the midwife after completion using study specific questionnaire.

   Adverse events/serious adverse events are documented and reported until 24 hours from completion of procedure.
4. Follow-up Further the questionnaire regarding patient experiences will be handed out one more time to the research person 24hours postpartum, or before discharge from hospital. Data from the patient's medical record will be extracted concerning pre-pregnancy-, pregnancy-and delivery data.

   Primary investigator may at any time withdraw a research person if the research person does not follow the procedures in the study protocol. Participation in the study is completely voluntary and the research subject may at any time terminate participation in the study without having to explain why and without incurring any consequences for further care. Upon termination of participation, treatment continues according to praxis on the clinic. Already collected data may be analysed if the research person does not oppose this.
5. End of trial The trial ends when the last subject has completed the last follow-up. Preliminary end of trial is set to the first half of 2024. The trial may be terminated prematurely if it proves necessary for safety reasons that affect the benefit/risk ratio or if the recruitment of test subjects cannot be fulfilled within reasonable time limits. If the trial is terminated prematurely, or temporarily stopped, the investigator must immediately inform the subjects of this and ensure appropriate treatment and follow-up. The Swedish Medical Products Agency should be informed via CTIS as soon as possible, but within 15 days at the latest. Decisions on early trial termination are made by the sponsor.

Presentation of the results are planned in regional, national, and international contexts, and the results will be sent for publication in an internationally recognized journal.

1. Selection of resarch subjects and Screening Patients that fulfil the inclusion criterions for the study will be given written and verbal information when admitted to the labor ward in active phase of labor. The patient is given verbal and written information about the study objectives, purpose and approach and will be given the opportunity to ask questions to the physician. After the delivery a check will be done if the patient still fulfils the inclusion criterions, and then the patient will again be given verbal and written information about the study objectives, purpose and approach and will be given the opportunity to ask questions to the physician before examination and repair of the perineal laceration. Participation is entirely voluntary. If the patient accepts study participation it results in a signed informed consent by the patient and physician before examination and repair of the perineal laceration. The recruitment to the study will be done by the physician. Patients, who fulfil the inclusion criteria will be recorded in a screening log. The informed consent form includes information that an independent monitor and medical regulatory authorities are allowed to compare data from the medical record with CRF. Reason for exclusion shall be documented in the log.
2. Criterions for cancellation of study The research person may cancel participation in the study at any time without having the further care affected.

   The sponsor/primary investigator may terminate the study prematurely if:
   * The participant does not follow the procedures in the study protocol.
   * Safety for the research persons within the study may be affected
   * Insufficient number of research persons can be included in the study
   * Study drugs according to the protocol cannot be delivered

   In case of a prematurely termination of study by the sponsor, this will be reported in CTIS to inform the Swedish MPA and EPM within 15 days together with a detailed written explanation of the reasons for termination.

   A research person is withdrawn from study by primary investigator if any of the following criteria are fulfilled:
   * research person withdrawal of informed consent
   * if research person safety is jeopardized
   * if the procedure is not possible to perform in accordance with the protocol due to insufficient sedation, insufficient pain relief or other circumstances.
3. Randomization The research subjects are included/randomized consecutively as they are deemed suitable to be included in the study.

There will be two arms: pudendal nerve block (group PNB) (todays standard of care) and pudendal nerve block with sedation using PCS with propofol (group PCS). The research subject will be randomized 1:1 to one of the two arms.

A sealed opaque randomization envelope containing instructions if PNB should be combined with PCS during the procedure. Randomization is done in blocks with equal distribution between the two groups. The envelopes for randomization are stored in a locked drug room at the clinic only accessible for staff at the clinic.

The research subject will be registered in a patient identification list with their personal identification number, full name and the assigned "Study ID".

Quality control and quality assurance

1. Department of Obstetrics and Gynaecology clinic at Vrinnevihospital in Norrköping Sweden, is the coordinating centre for the study with Linda Hjertberg as sponsor and primary investigator. The study team consists of the study actively participating researchers (physicians and midwifes).

   Before initiation of the study all concerned staff at the maternity ward will receive appropriate and customized education from anaesthetic staff regarding handling the patient-controlled device, pharmacological awareness of the IMP, routines, and practical training for emergency situations. The research team will provide detailed information for all staff involved in the study.

   The research team will have regular contact with the staff during the study period. Once the study is completed results of the study are presented to all personnel involved.

   The sponsor is responsible for implementing and maintaining quality assurance and quality control systems with written standard operating procedures to ensure that trials are conducted, and data are generated, documented, and reported in compliance with the protocol, ICH GCP, and Helsinki Declaration (2013).
2. Monitoring To ensure that the study is conducted according to the protocol, that data is collected, documented, and reported according to ICH-GCP as well as applicable ethical and regulatory requirements, the study will be monitored by an independent monitor before the start of the study, during the study and after the end of the study. The monitoring is carried out according to the study's monitoring plan and aims to ensure that the rights, safety, and well-being of the research subjects are met and that the data in the CRF is completed, correct and consistent with the source data.

   The investigator is obligated to give access to medical record for monitors, inspectors from the Swedish Medical Product Agency and any possible evaluators from the ethics committee.

   The monitor will ensure that informed consent is obtained according to regulations, compliance with the study protocol, to correct the data collected for the study developed CRF and that adverse events reported according to CTR 536/2014. Registration of the trial is done in CTIS in accordance with "The International Committee of Medical Journal Editors (ICMJE) Initiative" upon approval by the MPA and EPM.
3. Source data Source data is defined as any information in original records and certified copies of original records of clinical findings, observations or other activities necessary for reconstruction and evaluation for the study (e.g. CRF's, medical records). For this study, a separate Source Data Identification List will be written defining the source data for this study.
4. Deviations or serious violations Violations and deviations from trial protocols, GCP and other regulations that significantly directly affect, or with high probability would affect, research subjects in Sweden or the scientific value of the trial must be immediately reported by the sponsor within 7 days (from knowledge) to MPA through CTIS.

   Minor deviations that do not affect the integrity or safety of the research subjects, or significantly affect the scientific value of the trial, are documented in the trial documentation by the principal investigator and the sponsor.
5. Audit and inspections Authorized representatives of the sponsor and competent authorities may conduct audits or inspections at the trial site, including source data verification. The principal investigator must ensure that all source documents are available for audit and inspection. The purpose of an audit or inspection is to review all study-related activities and documents systematically and independently, to determine whether these activities were performed, recorded, analysed, and reported correctly according to the protocol, Good Clinical Practice (GCP) and applicable regulations.

Statistics

1. Sample size calculation A total of 70 research persons (35 research persons in each group) with a power of 80% and the investigators assume the overall statistically significant level for the trial is 0,05. To compensate for any dropouts or incomplete questionnaires the investigators add an additional 5 research persons to each group which results in 40 research persons in each group. Inclusion continues until 40 research persons in each group are included. The total study population will be 80 women.
2. Statistical method The primary outcome that are normally distributed will be analysed with Student's t-test. Secondary outcomes that are normally distributed will be analysed with Student's t-test else with the nonparametric test Mann-Whitney. Chi-squared test will be used for some of the secondary outcomes such as use of pain relief 24h postpartum to calculate difference between the expected frequencies. Safety variables with t-test or Mann-Whitney.
3. Dropouts and missing data Deviations from the study protocol will be treated individually. The CRF will be recorded midwife who individually will all have the right to make corrections of their individual records in the CRF. Data will be analysed according to intention-to-treat (ITT).

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥18 years)
* Planned examination and repair of perineal laceration
* The patient has after receiving verbal and written information about the study given her signed informed consent to participate

Exclusion Criteria:

* Perineal laceration grade III-IV
* BMI > 35 (during first visit at the maternity care centre)
* Deviation from department guidlines regarding preopartive fasting
* Preeclampsia or hypertensive disease
* Postpartum haemorrhage > 1000 ml
* Known/suspected allergy or contraindication to any medication within the study
* Functional disability in both hands which affect the possibility to operate the PCS device
* Cognitive impairment, unwillingness or language difficulties resulting in difficulty to understand the meaning of participation in the study or to operate the PCS device

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females after labor
Enrollment: 80 (Estimated)
Dates: Start 2023-09-20 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Pain/discomfort (perprocedural) | From randomization up to 2 hours. Measuring starts when the procedure with examination and repair of the laceration starts. Evaluation will be done immediately after procedure when criteria of fully recovered (OAA/S 5) is fulfilled.
  Perprocedural pain/discomfort; is a composite variable consisting measurements of pain and discomfort:
  Pain; measured with a VAS-scale (0-100 mm, "No pain" to "Worst imaginable pain") Discomfort; measured with a VAS-scale (0-100 mm, "No discomfort" to "Worst imaginable discomfort").

SECONDARY OUTCOMES:
Preprocedural anxiety | From randomization up to 2 hours. Evaluation will be done once in connection to completion of the procedure after fulfilling the criteria of fully recovered (OAA/S 5).
  Anxiety; measured with a VAS-scale (0-100 mm, "No anxiety" to "Worst imaginable anxiety").
Perprocedural anxiety | From randomization Up to 2 hours. Evaluation will be done once in connection to completion of the procedure after fulfilling the criteria of fully recovered (OAA/S 5).
  Anxiety; measured with a VAS-scale (0-100 mm, "No anxiety" to "Worst imaginable anxiety").
Patient experiences | From randomization Up to 2 hours. Evaluation will be done once in connection to completion of the procedure after fulfilling the criteria of fully recovered (OAA/S 5).
  Patient experiences (postprocedural) is measured using a study specific instrument.
Time of repair the perineal laceration | From randomization Up to 2 hours. Time for the procedure, the time between first attempt to suture until last suture.
  Time of repair the perineal laceration.
Ability to have skin-to-skin contact with baby during perineal repair | From randomization Up to 2 hours. The evaluation is made immediately after procedure completion.
  Ability to have skin-to-skin contact with baby during perineal repair; will recorded using a 4-point Likert scale with the items 1 (none), 2 (less than half of the procedure), 3 (more than half of the procedure) and 4 (during the whole procedure).
  Measured by the midwife.
Procedure feasibility (perprocedural) | From randomization Up to 2 hours.The evaluation is made immediately after procedure completion.
  Procedure feasibility (perprocedural) consists of several variables:
  Need of assistance from midwife; measured with a 3-items Likert scale (0="Not at all", 1="Partly", 2="Mostly") Need of assistance from partner; measured with a 3-items Likert scale (0="Not at all", 1="Partly", 2="Mostly", N/A) Ease of use; measured with a 4-items Likert scale (0="Easy", 1="Some difficulty", 2="Difficult", 3="Very difficult") Feasibility of PDB; 4-items Likert scale (0="Easy without any restrictions", 1="With somw difficulty but satisfactory result", 2="With som difficulty and impact on the result", 3="Had to cancel the procedure") Collaboration; measured with a 4-items Likert scale (0="None", 1="Minimal", 2="Moderate", 3="Significant") Defensive reactions/motions; measured with a 4-items Likert scale (0="None", 1="Minimal", 2="Moderate", 3="Significant") Overall satisfaction; measured with a 4-items Likert scale (0=" Satisfied", 1=" Neither satisfied nor dissatisfied/", 2=" Dissatisfied")
Amount of drugs used during perineal repair | From randomization Up to 2 hours. The evaluation is made immediately after procedure completion.
  Amount of drugs used during perineal repair; all drugs used during the procedure including PNB.
Time until micturition after the perineal repair | Time from randomization until 24 hours after. Evalutation time between completion of procedure until first in-ward micturition.
  Time until micturition after the perineal repair; is defined as time between completion of procedure until first in-ward micturition reported by the research person to staff.
Use of pain-relieving drugs 24h postpartum | On Day 1 after randomization. Evaluation after the first 24 hours after completion of procedure.
  Use of pain-relieving drugs 24h postpartum; type and amount of drugs for pain relief will be recorded for the first 24 hours after completion of procedure.
Patient experience | On Day 1 after randomization. Evaluates 24 hours after completion of procedure or upon discharge from hospital. Evalutation after 24 hours.
  Patient experience (at 24h postpartum or just before discharge from hospital with the same questions as asked directly after the procedure (OAA/S 5):
  Pain; measured with a VAS-scale (0-100 mm, "No pain" to "Worst imaginable pain").
  Discomfort; measured with a VAS-scale (0-100 mm, "No discomfort" to "Worst imaginable discomfort").
  Anxiety; measured with a VAS-scale (0-100 mm, "No anxiety" to "Worst imaginable anxiety").

OTHER OUTCOMES:
Peripheral capillary oxygen saturation | After randomization, From time to event. Recorded every five minutes during the procedure by monitoring oxygen saturation.
  Will be recorded Patient monitor Philips Intellivue MX700 and IntelliVue X3.
Respiratory frequency | After randomization,From time to event. Recorded every five minutes during the procedure by monitor Philips Intellivue MX700 and InterlliVueX3.
  Will be recorded Patient monitor Philips Intellivue MX700 and IntelliVue X3.
Non-invasive blood pressure | After randomization,From time to event. Recorded every five minutes during the procedure with monitor Philips Intellivue MX700 and IntelliVue X3.
  Will be recorded Patient monitor Philips Intellivue MX700 and IntelliVue X3.
Heart rate | After randomization,From time to event. Recorded every five minutes during the procedure with monitor Philips Intellivue MX700 and IntelliVue X3.
  Will be recorded Patient monitor Philips Intellivue MX700 and IntelliVue X3.
Level of sedation | After randomization,From time to event. Recorded every five minutes during the procedure
  Level of sedation; is assessed by the midwife using The Observer's Assessment of Alertness/Sedation (OAA/S) scale. The scoring of OAA/S scale specifying sedation level score between "Does not respond to mild prodding or shaking" (score 1) to "Responds readily to name spoken in normal tone" (score 5). Level of sedation is measured by the midwife in 5 minutes intervals until procedure completion.
Interventions | After randomization,From time of randomization to end of procedure with PNB or PNB+PCS.
  Interventions performed to maintain cardiovascular and respiratory stability; according to the pre-defined safety limits will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Hjertberg, MD, Principal Investigator — Department of Obstetrics and Gynecology, Vrinnevi Hospital, Sweden.
Locations (1):
- Vrinnevihospital, Norrköping, Sweden

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be available for sharing on request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The supporting information will be available from november 2025 until 6 months after publication
Access Criteria: Requests for sharing IPD that underlie results in a publication can be made to the principal investigator.